CLINICAL TRIAL: NCT01095185
Title: A Randomized, Multicenter,Double Blind,Controlled With Placebo Trial About Efficacy of Statin Association With Standard Treatment in Prevention of Recurrent Hemorrhage in Patient With Liver Cirrhosis and Variceal Bleeding
Brief Title: Efficacy of Statin Association With Standard Treatment in Prevention of Recurrent Hemorrhage in Patient With Cirrhosis and Variceal Bleeding
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Juan A. Arnaiz (Other)
Responsible Party: Sponsor-Investigator, Juan A. Arnaiz, Clinical Research Manager, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BLEPS; 2009-016500-24 (EudraCT Number)
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Cirrhosis; Hypertension, Portal; Bleeding Esophageal Varices; Portal Vein Thrombosis
MeSH Terms: conditions — Fibrosis; Hypertension, Portal | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard therapy + Simvastatin (Experimental): * Standard therapy: Endoscopic variceal ligation (EVL)+ B Blockers (Propanolol titrated until achieve maximum tolerated dose)
  * Simvastatin (20 mg for 15 days and after 40 mg/day until the end of the study)
  Interventions: Drug: Simvastatin
- Standard therapy + placebo (Placebo Comparator): * Standard therapy: Endoscopic variceal ligation (EVL)+ B Blockers (Propanolol titrated maximum tolerated dose).
  * Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 20 mg for 15 days, then 40 mg until the end of the study.
  Other Names: Simvastatina; Simvastatina Ratiopharm
  Arms: Standard therapy + Simvastatin
Drug: Placebo — Simvastatin placebo
  Arms: Standard therapy + placebo

SUMMARY:
This is a prospective, double blind controlled trial in which patients with esophagic variceal bleeding treated with standard therapy (endoscopic variceal ligation(EVL) + B-blockers), will be randomized to receive statins or placebo. They will be followed up during 12 months to determinate whether statins are effective in prevention of variceal bleeding recurrence and evaluate patient survival.

Randomization will be stratified according to the degree of hepatic insufficiency, assessed by the Child-Pugh classifications (A,B or C).

DETAILED DESCRIPTION:
A mayor cause of cirrhosis-related morbility and mortality is the development of variceal hemorrhage, a direct consequence of portal hypertension. In addition, survivors of an episode of active bleeding have a 70 % risk of recurrent hemorrhage within two years of the bleeding episode and the highest risk it is situated in the first six weeks after the hemorrhage episode.

The recommended treatment in AASLD guidelines is the combination of non selective Betablockers with endoscopic treatment with EVL, with high recurrence (30% in 2 years).

The hypothesis of this study is that statins are candidates for improving portal hypertension treatment in patients with cirrhosis, improving vascular function as well as preventing venous thrombotic events.

Patients with liver cirrhosis and variceal bleeding with standard treatment will be stratified and after randomized to undergo either statins (20 mg for 15 days, and after 40 mg/day) or placebo. They will be followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 80 years old.
* Clinical criteria and/or analytical, ultrasound and/or liver biopsy consistent with the diagnosis of liver cirrhosis.
* Hematemesis or melenas within 7 days prior to study inclusion.
* Variceal bleeding. Endoscopic diagnosis:

  * Active variceal bleeding.
  * Clot or platelet cluster or,
  * Esophageal varices associated to red blood in esophagogastric lumen in the absence of other sources of bleeding.
* Patients with standard treatment for prevention of recurrence of variceal bleeding (EVL+B Blockers,Propanolol).
* Women of childbearing age should have a urine pregnancy test negative for 7 days before commencement of treatment and postmenopausal women must have amenorrhea for at least 12 months to be considered not fertile. Potential childbearing women and men must commit to use adequate contraception prior to joining the study and during it.
* Written informed consent to participate in the study.

Exclusion Criteria:

* Pregnancy or lactation
* Presence multiple hepatocellular carcinoma or only diameter> 5 cm.
* Renal failure ( Creatinine > 2 mg/dl)
* Advanced liver disfunction (Child Pugh > 13 points)
* Contraindication for statins.
* Patients HIV treated with antiretroviral therapy.
* Pre-treatment with portosystemic shunt ( surgical or percutaneous).
* Bleeding due to gastric varices.
* Patients with total portal vein thrombosis or portal cavernomatosis.
* Patients previously treated with endoscopic variceal ligation and B- Blockers (before index episode).
* Patients previously treated with statins ( one month before the study).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Recurrence of variceal bleeding and patient survival | 12 months

SECONDARY OUTCOMES:
Bleeding severity in both arms. | 12 months
Appearance or progression of Portal Hypertension complications | 12 months
Appearance or progression of Portal Vein Thrombosis | 12 months
Need for alternative treatments (transjugular intrahepatic portosystemic shunt [TIPS], surgery) | 12 months
Incidence of adverse events of statin treatment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaume Bosch, MD, Principal Investigator — Hospital Clínic
Locations (15):
- Spain (15):
  - Hospital Universitario de Alicante, Alicante, Alicante
  - Hospital Clinic, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital German Trias i Pujol, Barcelona, Barcelona
  - Hospital de la Vall d'Hebron, Barcelona, Barcelona
  - Hospital Universitario del Mar, Barcelona, Barcelona
  - Hospital Universitari Bellvitge, L´Hospitalet Del LLobregat, Barcelona
  - Corporació Sanitària Parc Tauli, Sabadell, Barcelona
  - Hospital Arnau de Vilanova, Lleida, Catalonia
  - Complejo Hospitalario Pontevedra, Pontevedra, Galicia
  - Hospital Gregorio Marañon, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Puerta del Hierro, Majadahonda, Madrid
  - Complejo Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Tenerife

REFERENCES:
- [Derived] Abraldes JG, Villanueva C, Aracil C, Turnes J, Hernandez-Guerra M, Genesca J, Rodriguez M, Castellote J, Garcia-Pagan JC, Torres F, Calleja JL, Albillos A, Bosch J; BLEPS Study Group. Addition of Simvastatin to Standard Therapy for the Prevention of Variceal Rebleeding Does Not Reduce Rebleeding but Increases Survival in Patients With Cirrhosis. Gastroenterology. 2016 May;150(5):1160-1170.e3. doi: 10.1053/j.gastro.2016.01.004. Epub 2016 Jan 14. PMID 26774179